CLINICAL TRIAL: NCT03634228
Title: A Phase I/II Study of the Oral MDM2 Inhibitor DS-3032b (Milademetan) in Combination With Low Dose Cytarabine (LDAC) in Patients With Newly Diagnosed or Relapsed/Refractory Acute Myeloid Leukemia (AML)
Brief Title: Milademetan Tosylate and Low-Dose Cytarabine With or Without Venetoclax in Treating Participants With Recurrent or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to lack of adequate response, and did not move to the Phase II portion of the study
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0333; NCI-2018-01612 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0333 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (low dose cytarabine, MDM2 inhibitor DS-3032b) (Experimental): Patients receive low dose cytarabine SC BID on days 1-10 and milademetan tosylate PO QD on days 8-14, 8-21, or 5-7 and 15-17. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Milademetan Tosylate
- Phase II (low dose cytarabine, MDM2 inhibitor DS-3032b) (Experimental): Patients receive low dose cytarabine SC BID on days 1-10, milademetan tosylate PO QD on days 8-14, 8-21, or 5-7 and 15-17, and venetoclax PO QD on days 1-14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Milademetan Tosylate; Drug: Venetoclax

INTERVENTIONS:
Drug: Cytarabine — Given SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Milademetan Tosylate — Given PO
  Other Names: DS-3032 Tosylate; DS-3032b; DS-3032b Tosylate
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
  Arms: Phase II (low dose cytarabine, MDM2 inhibitor DS-3032b)

SUMMARY:
This phase I/II trial studies the side effects and best dose of milademetan tosylate and to see how well it works with cytarabine with or without ventoclax in treating participants with acute myeloid leukemia that has come back (recurrent) or that does not respond to treatment (refractory). Milademetan tosylate and ventoclax may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known if giving milademetan tosylate and low-dose cytarabine with or without ventoclax will work better in treating participants with recurrent or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study.

If you are enrolled in Phase 1, the dose of DS-3032b you receive will depend on when you join this study.

If you are enrolled in Phase 2, you will receive DS-3032b at the highest dose that was tolerated in Phase 1.

All participants will receive LDAC at a fixed dose (meaning the dose will not change). If you are assigned to receive it, your dose of venetoclax will not change either. However, if needed because you have side effects, your dose may be adjusted.

Up to 58 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) by World Health Organization (WHO) 2016 criteria. Patients will be divided into 2 arms during the phase 2 portion:

  * Arm A: Subjects must have newly diagnosed AML
  * Arm B: Subjects must have refractory or relapsed AML
* TP53 wild-type status on molecular testing performed within the last 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Creatinine clearance >= 60 mL/min, as calculated using the modified Cockcroft-Gault equation OR creatinine =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN
* Bilirubin =< 1.5 x ULN, unless resulting from hemolysis, Gilbert's disease or considered to be due to leukemic involvement
* No gastrointestinal issues to interfere with oral medication absorption
* No active uncontrolled infection or comorbidity that would interfere with therapy or place patient at increased risk
* Subject (male and female) of childbearing/reproductive potential must agree to use double-barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug
* Subject must sign and date an Institutional Review Board-approved informed consent form (including Health Insurance Portability and Accountability Act authorization, if applicable) before performance of any study-specific procedures or tests
* Able and willing to provide bone marrow biopsies/aspirates as requested by the protocol
* Willing to undergo malignancy genotyping for TP53 mutation, insertion, or deletion at screening
* Use of hydroxyurea is allowed prior to and during the first cycle of study treatment. 1-2 doses of cytarabine are also permitted if needed for cytoreduction prior to initiating study treatment

Exclusion Criteria:

* Patient with t(15;17) karyotypic abnormality or a diagnosis of acute promyelocytic leukemia
* Patient with other malignancy that contains a non-synonymous mutation, insertion, or deletion in the TP53 gene determined previously or at screening
* Prior treatment with an MDM2 inhibitor
* Presence of central nervous system involvement of leukemia. History of prior leptomeningeal leukemia/disease that has fully resolved is eligible
* A second concurrent primary malignancy that has required systemic anti-neoplastic treatment within the previous 6 months, except for localized cancers that have apparently been cured, for example non-melanoma skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast
* Any condition that would preclude adequate absorption of DS-3032b, including refractory vomiting, malabsorption, biliary shunt, significant bowel resection, and/or graft-versus-host disease (GVHD) affecting the gut
* Any active uncontrolled infection, known human immunodeficiency virus infection, or active hepatitis B or C infection
* Any concomitant medical condition that would in the opinion of the investigator increase the risk of toxicity
* Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5, grade =< 1 or baseline. Subjects with chronic grade 2 toxicities may be eligible per discretion of the investigator and sponsor (e.g., grade 2 chemotherapy-induced neuropathy)
* Patient having received hematopoietic stem cell transplantation (HSCT) within 60 days of the first dose of DS-3032b, is on immuno-suppressive therapy post-HSCT at the time of screening, or has clinically significant GVHD (use of topical steroids for ongoing skin GVHD will be permitted)
* Prolongation of corrected QT interval using Fridericia's method (QTcF) at rest, where the mean QTcF interval is >= 450 ms for males or >= 470 ms for females based on electrocardiograms (ECGs). Patients with right bundle branch block (RBBB) will be eligible after discussion with principal investigator (PI)
* Pregnant or breastfeeding
* Substance abuse or medical, psychological, or social conditions that, in the opinion of the investigator, may interfere with the subject's participation in the clinical study or evaluation of the clinical study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Senapati J, Muftuoglu M, Ishizawa J, Abbas HA, Loghavi S, Borthakur G, Yilmaz M, Issa GC, Dara SI, Basyal M, Li L, Naqvi K, Pourebrahim R, Jabbour EJ, Kornblau SM, Short NJ, Pemmaraju N, Garcia-Manero G, Ravandi F, Khoury J, Daver N, Kantarjian HM, Andreeff M, DiNardo CD. A Phase I study of Milademetan (DS3032b) in combination with low dose cytarabine with or without venetoclax in acute myeloid leukemia: Clinical safety, efficacy, and correlative analysis. Blood Cancer J. 2023 Jun 29;13(1):101. doi: 10.1038/s41408-023-00871-1. PMID 37386016
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0: Patients receive low dose cytarabine SC BID on days 1-10 and milademetan tosylate PO QD on days 8-14, 8-21, or 5-7 and 15-17. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cytarabine: Given SC
  Milademetan Tosylate: Given 120 mg PO
- Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1: Patients receive low dose cytarabine SC BID on days 1-10 and milademetan tosylate PO QD on days 8-14, 8-21, or 5-7 and 15-17. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cytarabine: Given SC
  Milademetan Tosylate: Given 200 mg PO
- Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2: Patients receive low dose cytarabine SC BID on days 1-10 and milademetan tosylate PO QD on days 8-14, 8-21, or 5-7 and 15-17. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cytarabine: Given SC
  Milademetan Tosylate: Given 260 mg PO
Period: Overall Study
Arm/Group | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2 | Phase II (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b)
Started | 3 | 6 | 7 | 0
Completed | 3 | 6 | 7 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2 | Total
Number analyzed (Participants) | 3 | 6 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 4 | 7
  >=65 years | 2 | 4 | 3 | 9
Age, Continuous [Median (Full Range); unit: years] | 72 [58 to 79] | 70 [38 to 77] | 53 [21 to 78] | 70 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 4 | 11
  Male | 2 | 0 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 2 | 4 | 5 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase I)
Description: As determined by dose limiting toxicity (DLT). MTD is defined the highest dose at which no more than one patient out of 6 patients experience DLTs in the first cycle. A 3+3 algorithm will be applied for dose escalation or dose de-escalation.
Time Frame: Up to 28 days
Measure: Number; unit: Milligrams
Arm/Group | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b)
Number analyzed (Participants) | 16
Milligrams | 260

2. Primary Outcome: Participants With a Response
Description: Response is Complete Response (CR) + Complete Response with Incomplete Blood Count Recovery (CRi) + Partial Response (PR) + Morphologic Leukemia -Free State (MLFS: CR is Bone marrow blasts < 5%; absence of circulating blasts and blasts with Auer rods; absence of extra-medullary disease; ANC >/= 1.0 x 10^9/L; platelet count >/= 100 x 10^9/L. CRi is CR except for ANC < 1.0 x 10^9 or platelet count , 100 x 10^9/L. PR is decreased bone marrow blast % by at least 50% to a value of 5% to 25% and ANC >/= 1.0 x 10^9/L; platelet count >/= 100 x 10^9/L. MLFS is Bone marrow blasts < 5%; abcence of blasts with Auer rods; absence of extra-medullary disease; no hematologic recovery required.
Time Frame: Up to 3 years, 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2
Number analyzed (Participants) | 3 | 6 | 7
Participants | 0 | 1 | 1

3. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 3 years, 4 months
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2
Number analyzed (Participants) | 3 | 6 | 7
Months | 2.1 [1.6 to 2.5] | 4.3 [0.6 to 28.4] | 7.6 [1.5 to 21.4]

4. Secondary Outcome: Event Free Survival (EFS)
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 3 years, 4 months
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2
Number analyzed (Participants) | 3 | 6 | 7
Months | 1.9 [1.6 to 2.5] | 2.4 [0.6 to 11.5] | 1.8 [1.4 to 7.3]

ADVERSE EVENTS:
Time Frame: Up to 3 years, 4 months
Arm/Group | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1 | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 7/7
Other Adverse Events (participants affected / at risk) | 2/3 | 0/6 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0 (N=3) | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1 (N=6) | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2 (N=7)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Eye Disorders (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 3 (4) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary Gland Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 4 (4) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 0 (N=3) | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 1 (N=6) | Phase I (Low Dose Cytarabine, MDM2 Inhibitor DS-3032b) Cohort 2 (N=7)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03634228/Prot_SAP_000.pdf